CLINICAL TRIAL: NCT05668416
Title: The Effect of Education Given to Parents of Children Undergoing Outpatient Surgery on Family-centered Care Perception and Anxiety: A Randomized Controlled Study
Brief Title: The Effect of Education Given to Parents of Children Undergoing Outpatient Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sevinc Akkoyun, lecturer (Phd), Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/46
Record Dates: First submitted 2022-12-03; First posted 2022-12-29 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Parents; Education; Children; Day Surgery; Family-centered Care; Anxiety
Keywords: Parents; education; children; day surgery; family-centered care; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial. In this parallel group study, intervention group and control group will take place.
Who Masked: Participant
Masking Description: Single (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment (Experimental): The intervention group will include parents who were trained in the preoperative period. The training includes brochures and oral training prepared by the researchers in line with the literature and the training given in the hospital.
  Interventions: Other: education
- control (No Intervention): The control group will be the oral information group that is in the hospital routine. Parents in this group will be informed verbally when they come to the hospital for anesthesia and file procedures the day before the surgery.

INTERVENTIONS:
Other: education — The training includes brochures and oral training prepared by the researchers in line with the literature and the training given in the hospital. Education brochure (Day surgery training brochure); An educational brochure was prepared by the researchers in line with the literature and practices in the institution. The brochure was composed of 3 sections: pre-operative, on the day of the operation and after the operation.
  Arms: experiment

SUMMARY:
The aim of the study is to examine the effect of the preoperative education given to the parents of the children who will undergo day surgery on the parents' perception of family-centered care and anxiety.

It is a randomized controlled trial. In this parallel group study, intervention group and control group will take place. The research will be carried out in the pediatric surgery service of the Selcuk University Medical Faculty Hospital. A total of 60 parents, including the intervention group (n=30) and the control group (n=30), will be included in the study. Parents to be included in the study will be assigned to intervention and control groups by randomization method. The randomization will be hidden from the researcher conducting the trial until the administration begins. The researcher will be given 60 envelopes and will begin to open the envelopes when he meets the parent. The researcher will learn which group each parent is in just before the application. Data collection tools; information form, state anxiety scale and Family Centered Care Assessment Scale. During the data collection phase, the purpose of the research will be explained to the parents by the researcher, information about the study will be given and consent will be obtained from the parents who agreed to participate in the research through the "Informed Voluntary Consent Form". A brochure prepared in line with the literature and the training given in the hospital will be given to the initiative group and verbal information will be given. On the other hand, only verbal information will be given to the control group, which is done in the hospital routine. The contents of the brochure include Preparation at Home 1 Day Before the Day of Surgery, Preparation at the Hospital on the Day of Surgery, and Home Care After the Surgery. Brochure and information will be given to the intervention group in the polyclinic one day before the surgery. Information Form, State Anxiety Scale and Family Centered Care Evaluation Scale will be filled in the polyclinic. The Information Form will be filled with the information obtained from the parents and the patient file. State Anxiety Scale and Family Centered Care Assessment Scale will be filled during discharge. Data will be analyzed with the IBM SPSS 22 (IBM Corporation, New York, NY) program. Partial eta squared will be calculated for the effect size and the significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
The aim of the study is to examine the effect of the preoperative education given to the parents of the children who will undergo day surgery on the parents' perception of family-centered care and anxiety.

It is a randomized controlled trial. In this parallel group study, intervention group and control group will take place. The research will be carried out in the pediatric surgery service of the Selcuk University Medical Faculty Hospital. The sample size of our study was determined by G-Power analysis. The analysis was determined as 24 parents (48 in total) in each group with 95% confidence interval, 0.05 margin of error, 1.08 effect size, 0.95 power. Data losses (25%) were also taken into account and 30 parents (60 in total) were determined for each group. Inclusion criteria; (a) Parents of children who had outpatient surgery, (b) Parents who can speak and understand Turkish, (c) Parents who volunteered to participate in the study. Exclusion criteria: (a) Parents of children who had elective surgery, (b) Parents of children who had previous surgery, (c) Parents with mental health problemsA total of 60 parents, including the intervention group (n=30) and the control group (n=30), will be included in the study. Parents to be included in the study will be assigned to intervention and control groups by randomization method. Control and intervention groups will be assigned by an independent statistician to reduce selection bias and control for variables that may affect the results. The randomization will be hidden from the researcher conducting the trial until the administration begins. The researcher will be given 60 envelopes and will begin to open the envelopes when he meets the parent. The researcher will learn which group each parent is in just before the application. Data collection tools; information form, state anxiety scale and Family Centered Care Assessment Scale. During the data collection phase, the purpose of the research will be explained to the parents by the researcher, information about the study will be given and consent will be obtained from the parents who agreed to participate in the research through the "Informed Voluntary Consent Form". A brochure prepared in line with the literature and the training given in the hospital will be given to the initiative group and verbal information will be given. On the other hand, only verbal information will be given to the control group, which is done in the hospital routine. The contents of the brochure include Preparation at Home 1 Day Before the Day of Surgery, Preparation at the Hospital on the Day of Surgery, and Home Care After the Surgery. Brochure and information will be given to the intervention group in the polyclinic one day before the surgery. Information Form, State Anxiety Scale and Family Centered Care Evaluation Scale will be filled in the polyclinic. The Information Form will be filled with the information obtained from the parents and the patient file. State Anxiety Scale and Family Centered Care Assessment Scale will be filled during discharge. Data will be analyzed with the IBM SPSS 22 (IBM Corporation, New York, NY) program. Partial eta squared will be calculated for the effect size and the significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with day surgery
* Parents who speak and understand Turkish
* Parents who volunteered to participate in the study

Exclusion Criteria:

* Parents of children who have had elective surgery
* Parents of children who have had previous surgery
* Parents with mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
anxiety level | 1 day before and after
  parents' anxiety levels
Perception of family-centered care level | 1 day before and after
  Parents' perception of family-centered care

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, professor, Study Director — Selcuk University; Tamer Sekmenli, associate professor, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The effect of the education given to the parents of the children who will undergo day surgery.
Supporting Information: Study Protocol
Time Frame: December 2022-March 2023 (3 months)

REFERENCES:
- [Derived] Akkoyun S, Arslan FT, Sekmenli T. The effect of written document in perioperative information on the anxiety level and family-centered care of parents of children undergoing ambulatory surgery: A randomized controlled trial. J Pediatr Nurs. 2024 Mar-Apr;75:108-115. doi: 10.1016/j.pedn.2023.12.012. Epub 2023 Dec 25. PMID 38147711